CLINICAL TRIAL: NCT02448654
Title: COMT Inhibition as a Novel Treatment for Nicotine Addiction in Women
Brief Title: Treatment for Nicotine Addiction in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1504015628; 1R21DA038253-01A1 (NIH)
Record Dates: First submitted 2015-05-14; First posted 2015-05-19 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tolcapone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolcapone (Active Comparator): 100mg tolcapone three times a day for 7 days then 100mg once a day on day 8
  Interventions: Drug: Sugar Pill
- Sugar Pill (Placebo Comparator): Sugar pill
  Interventions: Drug: Tolcapone

INTERVENTIONS:
Drug: Tolcapone — Tolcapone will be compared to sugar pill
  Other Names: Tasmar
  Arms: Sugar Pill
Drug: Sugar Pill — The sugar pill (placebo) will be compared to tolcapone
  Other Names: Placebo
  Arms: Tolcapone

SUMMARY:
The purpose of this study is to use a medication tolcapone and or placebo to test if the symptoms of nicotine withdrawal lessens , and or changes in smoking urges, and mental reasoning in female smokers over a 72 hour period.

DETAILED DESCRIPTION:
The proposed trail will be use a double-blind, placebo-controlled design to conduct the first randomized controlled trial of the COMT inhibitor, tolcapone, in nicotine dependent women. This study will determine if tolcapone is superior to placebo by attenuation the severity of nicotine withdrawal and smoking urges during short-term abstinence. Withdrawal severity will be assessed by a self-report scale and cognitive assessment, including a sustained-attention task. Smoking urges will be assessed by a self-report scale.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18yrs to 45yr old woman, read and write in English.
* Must smoke at least 5 or more cigarettes a day
* FTND score at least 4 or higher
* A CO reading of 10 or higher during screening
* Must be in good health as verified by medical history, screening exam, screen laboratory tests.

Exclusion Criteria:

* Excluded if using psychotropic medications, have contraindications to tolcapone use (e.g.. liver problems, allergy to tolcapone, history of no traumatic rhabdomyolysis or hyperpyrexia, confusion possibly related to medication), have other substance use disorder, are pregnant or breast feeding, have a current psychotic disorder, bipolar disorder, homicidal or suicidal ideation, have current (past month) substance use disorder, other than nicotine dependence, or are unable to fulfill the scheduled visits and procedures.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elise DeVito, Ph.D., Principal Investigator — Yale University
Locations (1):
- Veterans Administration Hospital, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 36 consented to be in the study, completed a baseline session, and were randomized to a study arm. However, 4 subjects never actually began the medication trial (i.e., stopped participating prior to receiving any pills (tolcapone or placebo)). 32 subjects began the pill portion of the trial (i.e., started tolcapone or placebo).
Groups:
- Sugar Pill: Sugar pill (placebo) three times a day for 7 days then once on day 8
Period: Overall Study
Arm/Group | Tolcapone | Sugar Pill
Started (Were eligible and completed the baseline assessments.) | 19 | 17
Started Pills (Tolcapone or Placebo) (Started the medication (tolcapone or placebo) portion of the trial.) | 17 | 15
Completed (Completed the medication (tolcapone or placebo) trial.) | 16 | 13
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Population: Eligible and completed baseline assessment
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolcapone | Sugar Pill | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.16 (7.88) | 33.35 (7.77) | 32.72 (7.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 17 | 13 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 14 | 7 | 21
  White | 2 | 10 | 12
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Withdrawal Symptoms (MNWS Score)
Description: The MNWS was the 8 item version, using VAS scales for each item (1-100), and MNWS score calculated as an average of all items (range of possible scores for MWNS at each timepoint was 0-100, with higher MNWS scores at each timepoint indicating more withdrawal symptoms (worse outcome). Timepoints reflect 1.) the baseline (beginning of the trial, not yet receiving any pills, not yet being asked to abstain from smoking; calculated as average of scores from two visits: ad libitum baseline visit and pill day 1 measure which was collected prior to administration of pills) and 2.) the abstinence period (tolcapone or placebo pill days 6-8, during the 60-hr abstinence phase; calculated as average of scores from 3 visits: pill days 6, 7, and 8). Greater increases in scores (increases in withdrawal symptoms) during abstinence period compared to baseline reflects a worse outcome; reduced or stable scores (decreases or a lack of increases in withdrawal symptoms) during the abstinence period compa
Time Frame: Baseline (ad libitum baseline and pill day 1 (pre-pill)); Abstinent Period (pill days 6, 7, 8)
Population: Study completers (participants who were eligible, randomized to a treatment condition, and completed the study).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tolcapone | Sugar Pill
Number analyzed (Participants) | 16 | 13
score on a scale
  Baseline (no pills, not abstinent) | 13.33 (8.48) | 9.40 (8.12)
  Abstinent Period (on pills, nicotine abstinent)) | 11.95 (11.80) | 13.29 (13.07)
Statistical Analysis 1: Comparison: Tolcapone vs Sugar Pill; Test type: Superiority; p = 0.18, ANOVA — The a priori threshold for statistical significance was p<0.05

2. Primary Outcome: Smoking Urges (BQSU Factor 1)
Description: The Brief Questionnaire on Smoking Urges (BQSU) is a 10 item scale. Factor 1 reflects the urge to smoke for its rewarding properties. Factor 1 is calculated as the sum of five items (items 1, 3, 6, 7, 10), with each item score ranging from 1-7, so Factor 1 scores range from 5-35. Higher scores reflect higher smoking urges and represent a worse outcome. Timepoints reflect 1.) baseline (beginning of trial, not yet receiving pills, not yet abstaining from smoking; calculated as average of scores from ad libitum baseline visit and pill day 1 which was collected prior to administration of pills) and 2.) abstinence period (pill days 6-8, during 60-hr abstinence phase; calculated as average of scores from pill days 6, 7, and 8). Greater increases in scores (increases in smoking urges) during abstinence period compared to baseline reflects a worse outcome; decreases or a lack of increases in smoking urges during the abstinence period compared to baseline reflects a better outcome.
Time Frame: Baseline (ad libitum baseline and pill day 1 (pre-pill)); Abstinent Period (pill days 6, 7, 8)
Population: Study completers (participants who were eligible, randomized to a treatment condition, and completed the study).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tolcapone | Sugar Pill
Number analyzed (Participants) | 16 | 13
score on a scale
  Baseline (no pills, not abstinent) | 19.69 (9.89) | 13.42 (7.44)
  Abstinent Period (on pills, nicotine abstinent)) | 14.50 (10.42) | 16.04 (9.58)
Statistical Analysis 1: Comparison: Tolcapone vs Sugar Pill; Test type: Superiority; p = 0.03, ANOVA — The a priori threshold for statistical significance was p<0.05

3. Primary Outcome: Smoking Choice Paradigm: Amount Earned ($)
Description: The Smoking Choice Paradigm was done once at the end of the trial (Pill Day 8, at the end of the 60 hr abstinence period). Subjects are given forced choice options between 2 puffs of their own-brand cigarette vs. a token with a monetary value, spaced over a 90 minute period. The maximum amount subjects can earn from this task ranges from $0 to $7.50 (10 forced choice opportunities: smoke 2 puffs vs. earn 75 cent at each choice opportunity). Higher earnings reflect choice of the tokens over smoking, so this reflects a better outcome (i.e., reduced smoking choice).
Time Frame: Pill-Day 8 (end of trial)
Population: Study completers (participants who were eligible, randomized to a treatment condition, and completed the study).
Measure: Mean (Standard Deviation); unit: Dollars ($)
Arm/Group | Tolcapone | Sugar Pill
Number analyzed (Participants) | 16 | 13
Dollars ($) | 7.41 (0.26) | 7.06 (0.57)
Statistical Analysis 1: Comparison: Tolcapone vs Sugar Pill; Test type: Superiority; p = 0.037, ANOVA — The a priori threshold for statistical significance was p<0.05

ADVERSE EVENTS:
Time Frame: During the medication phase (8 days) and follow-up (1 week).
Description: Patients 'at risk' for all adverse events are the 'safety population'- which consists of any patient that received study drug post randomization. This would be a total of 32 of 36 patients, 17 in Tolcapone arm and 15 in Sugar Pill arm.
Arm/Group | Tolcapone | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 12/17 | 14/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolcapone (N=17) | Sugar Pill (N=15)
Stomach pain (Gastrointestinal disorders) | 3 (4) | 1 (1)
Upset stomach (Gastrointestinal disorders) | 1 (2) | 4 (6)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1)
Loss of appetite (Gastrointestinal disorders) | 2 (3) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Nervousness (Psychiatric disorders) | 0 (0) | 5 (9)
Restlessness (Psychiatric disorders) | 2 (2) | 7 (12)
Difficulty sleeping (Psychiatric disorders) | 3 (3) | 9 (12)
Feeling drowsy (Psychiatric disorders) | 5 (6) | 5 (9)
Extreme tiredness (fatigue) (Psychiatric disorders) | 5 (6) | 3 (4)
Anger or irritability (Psychiatric disorders) | 1 (2) | 5 (10)
Depressed mood (Psychiatric disorders) | 1 (2) | 4 (11)
Teary or dry eyes (Eye disorders) | 2 (2) | 2 (11)
Nosebleed (General disorders) | 1 (1) | 1 (1)
Runny nose (General disorders) | 0 (0) | 4 (5)
Back muscle or bone pain (Musculoskeletal and connective tissue disorders) | 5 (9) | 3 (7)
Sweating (General disorders) | 2 (3) | 1 (1)
Rash or skin problem (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (11)
Excessive Hunger (Gastrointestinal disorders) | 4 (4) | 3 (6)
Inability to respond to things around you (Psychiatric disorders) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 3 (4) | 3 (4)
Change in ability to taste food (Gastrointestinal disorders) | 2 (4) | 2 (2)
Headache (Psychiatric disorders) | 3 (3) | 10 (12)
Tremors or shakiness (General disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Slowed thinking (Psychiatric disorders) | 1 (1) | 0 (0)
Tingling in fingers or toes (General disorders) | 3 (6) | 1 (1)
Sore Throat (General disorders) | 2 (3) | 3 (7)
Fever (General disorders) | 1 (1) | 2 (3)
Chills (General disorders) | 2 (4) | 2 (2)
Slow heart rate (Cardiac disorders) | 1 (1) | 0 (0)
Crossed eyes (Eye disorders) | 2 (4) | 1 (1)
Gas (Gastrointestinal disorders) | 3 (5) | 3 (8)
Irregular or pounding heartbeat (Cardiac disorders) | 2 (2) | 1 (1)
Feeling dizzy or faint or lighheaded (General disorders) | 2 (3) | 3 (4)
Weightloss (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Eye pain (Eye disorders) | 1 (2) | 0 (0)
Numbness or tingling around mouth (General disorders) | 1 (2) | 0 (0)
Problems with urination (Renal and urinary disorders) | 1 (1) | 0 (0)
Slowed movements (General disorders) | 1 (2) | 0 (0)
Sudden hunger (General disorders) | 3 (4) | 1 (3)
Trouble speaking or swallowing (General disorders) | 1 (1) | 0 (0)
Difficulty concentrating (Psychiatric disorders) | 1 (2) | 1 (5)
Memory problems (Psychiatric disorders) | 2 (2) | 1 (5)
Seizures (Psychiatric disorders) | 1 (1) | 0 (0)
Swelling of tongue (General disorders) | 1 (1) | 0 (0)
Trouble with gums (General disorders) | 1 (1) | 1 (1)
Extreme thirst (General disorders) | 1 (1) | 2 (2)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Aggressive behavior (Psychiatric disorders) | 2 (3) | 1 (1)
Mood swings (Psychiatric disorders) | 2 (2) | 4 (4)
Dandruff (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (8)
Growth of hair in unusual places (Endocrine disorders) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Trouble walking (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Kidney Stones (Renal and urinary disorders) | 1 (1) | 0 (0)
Involuntary eye movements (Eye disorders) | 1 (2) | 0 (0)
Near Sightedness (Eye disorders) | 2 (3) | 0 (0)
Breast pain (female only) (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Painful menstrual periods (female only) (Reproductive system and breast disorders) | 2 (3) | 2 (7)
Missed menstrual periods (female only) (Reproductive system and breast disorders) | 2 (3) | 1 (5)
Excessive Menstrual Bleeding (female only) (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/54/NCT02448654/Prot_000.pdf
  • Statistical Analysis Plan (2014-07-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT02448654/SAP_001.pdf